CLINICAL TRIAL: NCT06332196
Title: Immunodeficiency and Cancer: Identification of Congenital Immune System Defects Underlying Paediatric Lymphomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Eleonora Gambineri, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: L-IEI
Record Dates: First submitted 2024-02-24; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Immune Deficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with non-Hodgkin's lymphoma (NHL) or Hodgkin's lymphoma (HL) aged and patients with previous lymphoma and signs of immunodeficiency
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Hodgkin's lymphoma (HL) or non-Hodgkin's lymphoma (NEIL) (Other): Patient with Hodgkin's lymphoma (HL) or non-Hodgkin's lymphoma (NEIL)
  Interventions: Other: Analysis of biological sample and clinical data

INTERVENTIONS:
Other: Analysis of biological sample and clinical data — Analysis of biological sample and clinical data

SUMMARY:
Inborn Errors of Immunity (IEI) are a heterogeneous group of disorders characterised not only by an infectious diathesis, but by a wide variety of other clinical manifestations. Lymphoma is one of the most common malignancies in children and may be the first clinical manifestation of IEI, thereby 'hiding' the immune defect and delaying genetic/immunological diagnosis. Lymphomas, especially non-Hodgkin's lymphomas (NHL) are frequently associated with congenital defects of the immune system, in particular diffuse large B-cell lymphoma and Burkitt's lymphoma. Preliminary analyses conducted on 6 patients diagnosed with NHL allowed the identification of genetic variants in genes associated with IEI. In clinical practice, the diagnosis and choice of therapeutic treatment in patients with immunodeficiency-associated lymphoma are decisive and, due to the complex pathophysiology of the disease, it is not always possible to identify the boundary between benign and malignant proliferation. The identification of an undiagnosed immunodeficiency in patients with lymphoma will ensure the opportunity to apply targeted therapies, such as allogeneic haematopoietic stem cell transplantation, instead of standard clinical management based mainly on chemotherapy. The study aims to identify possible congenital defects of immunity, i.e. genetic disorders affecting the immune system, as responsible for the development of haematological malignancies. Through a multidisciplinary approach involving immunological analyses, genetic analyses and a thorough examination of clinical manifestations, we aim to characterise the immunological component underlying the development of paediatric lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of Hodgkin's lymphoma (HL) or non-Hodgkin's lymphoma (NEIL) with or without signs of immune dysregulation (lymphoproliferation, autoimmunity, hypogammaglobulinaemia, family history of immunodeficiency).
* Patients with previous HL or NEIL lymphoma who have developed, concomitantly with the tumour or subsequently, clinical manifestations mentioned above attributable to a congenital defect of immunity.

Exclusion Criteria:

* Patients with known genetic diseases, or who do not consent to participate in the study

Ages: 1 Day to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-06-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
To unravel inborn error of immunity behind Lymphoid neoplasm in children | Through study completion, an average of 1 year
  Characterizing the role of the immune system in the pathogenesis of polyclonal and clonal lymphoproliferation. In particular, the main aim of our study will be the identification, by means of second-generation genetic analysis and functional validation studies of the identified variants, of congenital immune system defects in patients with lymphoid neoplasia

SECONDARY OUTCOMES:
Identification of lymphoma-specific biomarkers | Through study completion, an average of 1 year
  Investigating Cell-Free DNA for specific molecular alterations in lymphomas, in order to monitor the follow-up of patients affected by lymphoma and to identify early onset of clonality in patients with already diagnosed congenital defects of the immune system at risk of developing malignant lymphoproliferation.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Gambineri, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (4):
- Italy (4):
  - AOU Malpighi IRCCS, Bologna
  - Meyer Children's Hospital IRCCS, Florence
  - AOU Pisana, Pisa
  - Ospedale Pediatrico Bambin Gesù IRCCS, Roma